CLINICAL TRIAL: NCT04574752
Title: MSSA and MRSA Screening in Patients Undergoing Elective TJA: the Benefits of Next-generation Sequencing
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Other Study IDs: JPARV20D.165
Record Dates: First submitted 2020-09-29; First posted 2020-10-05 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: Staphylococcus Aureus; Next Generation Sequencing; Total Joint Arthroplasty
MeSH Terms: conditions — Staphylococcal Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: next generation sequencing — diagnostic performance of molecular and culture techniques in S. aureus screening using paired nasal and groin swabs, to determine, if any, discrepancy between the diagnostic techniques on S. aureus detection in orthopaedic patients

SUMMARY:
The aims of this study were to evaluate the diagnostic performance of molecular and culture techniques in S. aureus screening using paired nasal and groin swabs, to determine, if any, discrepancy between the diagnostic techniques and to model the potential effect of different diagnostic techniques on S. aureus detection in orthopaedic patients

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing primary total knee or total hip arthroplasty at our institution will be eligible.

Exclusion Criteria:

* Patients included in other prospective studies

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients undergoing primary total knee or total hip arthroplasty at our institution will be eligible
Sampling Method: Non-Probability Sample
Enrollment: 163 (Actual)
Dates: Start 2020-08-30 (Actual); Primary Completion 2021-08-30 (Estimated); Study Completion 2021-08-30 (Estimated)

PRIMARY OUTCOMES:
Diagnostic techniques to identify S. aureus in total joint replacement patients | 1 day
  to model the potential effect of different diagnostic techniques on S. aureus detection in orthopaedic patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Rothman Orthopaedic Institute, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No